CLINICAL TRIAL: NCT05165485
Title: A Phase 4, Randomized, Double-Blind, Double-Dummy, Parallel-Group, Study Comparing Improvements in Lung Function in Adults With Severe to Very Severe Chronic Obstructive Pulmonary Disease and Suboptimal Inspiratory Flow Rate Following Once-Daily Treatment Over 12 Weeks With Either Revefenacin Inhalation Solution Delivered Via Standard Jet Nebulizer or Tiotropium Delivered Via a Dry Powder Inhaler (Spiriva® HandiHaler®)
Brief Title: Phase 4 COPD and Suboptimal Inspiratory Flow Rate
Acronym: PIFR-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Collaborators: Viatris Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0180
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Peak Inspiratory Flow Rate; PIFR; Pulmonary Function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — revefenacin; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Revefenacin (Experimental): Revefenacin administered with Tiotropium Placebo
  Interventions: Drug: Revefenacin; Drug: Tiotropium Placebo
- Tiotropium (Active Comparator): Tiotropium administered with Revefenacin Placebo
  Interventions: Drug: Tiotropium; Drug: Revefenacin Placebo

INTERVENTIONS:
Drug: Revefenacin — Revefenacin 175 mcg administered once daily for 84 days via nebulization
  Other Names: Yupelri®; TD-4208
  Arms: Revefenacin
Drug: Tiotropium — Tiotropium 18 mcg administered once daily for 84 days via Spiriva HandiHaler®
  Other Names: Spiriva®
  Arms: Tiotropium
Drug: Revefenacin Placebo — Placebo for Revefenacin administered once daily for 84 days via nebulization
  Arms: Tiotropium
Drug: Tiotropium Placebo — Placebo for Tiotropium administered once daily for 84 days via Spiriva HandiHaler®
  Arms: Revefenacin

SUMMARY:
Study is a randomized, double-blind, double-dummy, parallel-group study evaluating efficacy and safety of revefenacin vs. tiotropium in adults with severe to very severe COPD and suboptimal PIFR.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is a male or female 40 years of age or older.
2. Participant is female and is nonpregnant and nonlactating. A woman of childbearing potential must have a documented negative urine pregnancy test at screening. Women are considered not to be of childbearing potential if they have had a total hysterectomy and/or bilateral tubal ligation (documentation for either must be provided before enrollment) or are at least 2 years postmenopausal.
3. During the study and for 30 days after receiving the last dose of study drug, women of childbearing potential and men capable of fathering children must agree to use highly effective birth control measures or agree to abstain from sexual intercourse.

   A highly effective method of birth control is defined as one that results in a low failure rate (i.e. <1% per year) when used consistently and correctly, such as condom + diaphragm, condom + spermicide, diaphragm + spermicide, or intrauterine device [IUD] with documented failure rate of <1% per year, or oral/injectable/implanted hormonal contraceptives used in combination with an additional barrier method.
4. Participant has a diagnosis of COPD, specifically, a post-ipratropium FEV1/FVC ratio <0.7.
5. Participant has a post ipratropium 30% ≤ FEV1 < 50% of predicted normal (using National Health and Nutrition Examination Survey-predicted equations) and absolute FEV1 > 500 mL, or FEV1 <30% predicted normal and absolute FEV1 > 700 mL.
6. Participant has a PIFR <60 L/min as measured by an In-Check™ device with resistance set to DISKUS at Visit 1A (if not combined with Visit 1B) and < 55 L/min as measured by an In-Check™ device with resistance set to DISKUS at Visit 1B and Visit 2 prior to randomization.
7. Participant is capable of performing reproducible spirometry maneuvers (and plethysmography maneuvers for a subset of participants) as described by current American Thoracic Society (ATS) Guidelines.
8. Participant is an active or former smoker with a cigarette smoking history (or equivalent for cigar or pipe smoking history) of at least 10 pack-years.
9. Participant or legal guardian is willing and able to provide signed and dated informed consent to participate prior to initiation of any study related procedures.
10. Participant is willing and able to adhere to all study assessments/procedures. Care partner assistance is acceptable.
11. Participant is willing and able to adhere to all restrictions during their study participation as follows:

    * Use of recreational drugs
    * Medicinal marijuana
    * Excessive alcohol during the study period
    * Participation in another investigational drug study
    * Donation of ≥500 mL blood (or equivalent)
12. Participant (or care partner) based on the investigator's assessment is able to properly prepare and administer study medication administered from both nebulizer and HandiHaler® according to their respective Instructions for Use.

Exclusion Criteria:

1. Participant has a concurrent disease or condition that, in the opinion of the investigator, would interfere with study participation or confound the evaluation of safety and tolerability of the study drug.
2. Participant has a history of reactions or hypersensitivity to inhaled or nebulized anticholinergics.
3. Participant suffers from any medical condition that would preclude the use of inhaled anticholinergics, including narrow-angle glaucoma, symptomatic benign prostatic hyperplasia, bladder neck obstruction, or urinary retention.
4. Participant has Moderate to Severe Hepatic impairment (Child-Pugh B or C) or Severe Renal Insufficiency (i.e. a glomerular filtration rate <30 mL/min/1.72m^2).
5. Participant has been hospitalized for COPD or pneumonia within 8 weeks prior to Visit 1.
6. Participant is receiving a LABA or LABA/inhaled corticosteroid (ICS; either QD or BID) at a dose that has been stable for ≤ 30 days prior to screening.
7. Participant has used systemic corticosteroids within 8 weeks of Visit 1.
8. Participant has used antibiotics for respiratory tract infections within 8 weeks of Visit 1, or is using antibiotics prophylactically.
9. Participant received COVID-19 vaccine within 2 weeks prior to Visit 1.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (72):
- United States (72):
  - Theravance Biopharma Investigational Site, Jasper, Alabama
  - Theravance Biopharma Investigational Site, Phoenix, Arizona
  - Theravance Biopharma Investigational Site, Tucson, Arizona
  - Theravance Biopharma Investigational Site, Newport Beach, California
  - Theravance Biopharma Investigational Site, San Diego, California
  - Theravance Biopharma Investigational Site, Stockton, California
  - Theravance Biopharma Investigational Site, Upland, California
  - Theravance Biopharma Investigational Site, Lakewood, Colorado
  - Theravance Biopharma Investigational Site, Brandon, Florida
  - Theravance Biopharma Investigational Site, Clearwater, Florida
  - Theravance Biopharma Investigational Site site 2, Clearwater, Florida
  - Theravance Biopharma Investigational Site, Daytona Beach, Florida
  - Theravance Biopharma Investigational Site, Leesburg, Florida
  - Theravance Biopharma Investigational Site, Miami, Florida
  - Theravance Biopharma Investigational Site, Orlando, Florida
  - Theravance Biopharma Investigational Site, Ormond Beach, Florida
  - Theravance Biopharma Investigational Site, Sarasota, Florida
  - Theravance Biopharma Investigational Site, Tampa, Florida
  - Theravance Biopharma Investigational Site, Winter Park, Florida
  - Theravance Biopharma Investigational Site, Chicago Ridge, Illinois
  - Theravance Biopharma Investigational Site, River Forest, Illinois
  - Theravance Biopharma Investigational Site, Hammond, Indiana
  - Theravance Biopharma Investigational Site, Valparaiso, Indiana
  - Theravance Biopharma Investigational Site, Annapolis, Maryland
  - Theravance Biopharma Investigational Site, Columbia, Maryland
  - Theravance Biopharma Investigational Site, Oxon Hill, Maryland
  - Theravance Biopharma Investigational Site, Towson, Maryland
  - Theravance Biopharma Investigational Site, North Dartmouth, Massachusetts
  - Theravance Biopharma Investigational Site, Farmington Hills, Michigan
  - Theravance Biopharma Investigational Site, Saint Charles, Missouri
  - Theravance Biopharma Investigational Site, St Louis, Missouri
  - Theravance Biopharma Investigational Site, Missoula, Montana
  - Theravance Biopharma Investigational Site, Las Vegas, Nevada
  - Theravance Biopharma Investigational Site, Albuquerque, New Mexico
  - Theravance Biopharma Investigational Site, Bronxville, New York
  - Theravance Biopharma Investigational Site, Schenectady, New York
  - Theravance Biopharma Investigational Site, Charlotte, North Carolina
  - Theravance Biopharma Investigational Site, Hickory, North Carolina
  - Theravance Biopharma Investigational Site, Huntersville, North Carolina
  - Theravance Biopharma Investigational Site, Kernersville, North Carolina
  - Theravance Biopharma Investigational Site, Monroe, North Carolina
  - Theravance Biopharma Investigational Site, Raleigh, North Carolina
  - Theravance Biopharma Investigational Site, Winston-Salem, North Carolina
  - Theravance Biopharma Investigational Site, Cincinnati, Ohio
  - Theravance Biopharma Investigational Site, Columbus, Ohio
  - Theravance Biopharma Investigational Site, Marion, Ohio
  - Theravance Biopharma Investigational Site, Grants Pass, Oregon
  - Theravance Biopharma Investigational Site, Medford, Oregon
  - Theravance Biopharma Investigational Site, Portland, Oregon
  - Theravance Biopharma Investigational Site, Anderson, South Carolina
  - Theravance Biopharma Investigational Site, Columbia, South Carolina
  - Theravance Biopharma Investigational Site, Gaffney, South Carolina
  - Theravance Biopharma Investigational Site, Greenville, South Carolina
  - Theravance Biopharma Investigational Site, Lexington, South Carolina
  - Theravance Biopharma Investigational Site, North Charleston, South Carolina
  - Theravance Biopharma Investigational Site, Rock Hill, South Carolina
  - Theravance Biopharma Investigational Site #2, Spartanburg, South Carolina
  - Theravance Biopharma Investigational Site, Spartanburg, South Carolina
  - Theravance Biopharma Investigational Site, Union, South Carolina
  - Theravance Biopharma Investigational Site, Franklin, Tennessee
  - Theravance Biopharma Investigational Site, Johnson City, Tennessee
  - Theravance Biopharma Investigational Site, Knoxville, Tennessee
  - Theravance Biopharma Investigational Site, Kerrville, Texas
  - Theravance Biopharma Investigational Site, McAllen, Texas
  - Theravance Biopharma Investigational Site, San Antonio, Texas
  - Theravance Biopharma Investigational Site, Sherman, Texas
  - Theravance Biopharma Investigational Site, Webster, Texas
  - Theravance Biopharma Investigational Site, Roy, Utah
  - Theravance Biopharma Investigational Site, West Valley City, Utah
  - Theravance Biopharma Investigational Site, Abingdon, Virginia
  - Theravance Biopharma Investigational Site, Spokane, Washington
  - Theravance Biopharma Investigational Site, Cudahy, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

RESULTS

PARTICIPANT FLOW:
Groups:
- Tiotropium: Active Tiotropium and Placebo for Revefenacin.
  Tiotropium: Tiotropium administered via Spiriva HandiHaler® device. Placebo for Revefenacin: Placebo administered as double blind, double dummy via nebulization.
- Revefenacin: Active Revefenacin and Placebo for Tiotropium.
  Revefenacin: Revefenacin administered via nebulization. Placebo for Tiotropium: Placebo administered as double blind, double dummy via HandiHaler® device.
Period: Overall Study
Arm/Group | Tiotropium | Revefenacin
Started (A total of 23 enrolled participants from 2 sites are excluded from the Participant Flow table and all analysis populations due to data integrity concerns.) | 191 | 190 (A total of 190 participants were randomized to the Revefenacin group and 189 received study treatment. One participant did not start study treatment.)
Completed | 156 | 147
Not Completed | 35 | 43

BASELINE CHARACTERISTICS:
Population: All participants who received study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium | Revefenacin | Total
Number analyzed (Participants) | 191 | 189 | 380
Age, Continuous [Median (Full Range); unit: years] | 66 [49 to 88] | 67 [47 to 83] | 66 [47 to 88]
Age, Customized [Count of Participants; unit: Participants]
  40 to 64 years old | 81 | 79 | 160
  65 years old and over | 110 | 110 | 220
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 90 | 176
  Male | 105 | 99 | 204
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 176 | 172 | 348
  Unknown or Not Reported | 13 | 10 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 11 | 14 | 25
  White | 175 | 171 | 346
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 191 | 189 | 380

OUTCOME MEASURES:

1. Primary Outcome: FEV1
Description: Change from baseline in forced expiratory volume in one second (FEV1) at trough on Day 85
Time Frame: Baseline, Day 85 following 84 days of dosing
Population: All participants who received study treatment
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Tiotropium | Revefenacin
Number analyzed (Participants) | 191 | 189
mL | 101 (17) | 78 (17)
Statistical Analysis 1: Comparison: Tiotropium vs Revefenacin; The null hypothesis was that the Revefenacin - Tiotropium Least Squares Mean Difference was zero and the alternative hypothesis was that it was nonzero; Test type: Superiority; p = 0.22, Mixed Models Analysis — The familywise type 1 error rate is controlled at 0.05 by testing the primary and secondary endpoint hypotheses in sequence, stopping after the first failure to reject the null hypothesis; Denominator degrees of freedom were approximated by the Kenward and Roger (1997) method; Mean Difference (Net) = -23, 95% CI 2-sided [-61 to 14] — Revefenacin - Tiotropium Least Squares Mean Difference; The Revefenacin - Tiotropium Least Squares Mean Difference was estimated by fitting a repeated measures mixed model which included terms for participant, treatment, 6 categorical covariates, and 3 continuous covariates: baseline FEV1, screening FEV1, and baseline PIFR. The 6 categorical covariates were reversibility to ipratropium status (reversible/not reversible), smoking status (current/former), concomitant LABA or LABA/ICS use (Yes/No), GOLD airflow category (3/4, i.e., postipratropium FEV1 % predicted < 30%/≥ 30%), sex (woman/man), and age group (< 65/≥ 65)

2. Secondary Outcome: OTE on FEV1
Description: Trough Overall Treatment Effect (OTE) on FEV1. Overall is defined as the average change from baseline at trough across Day 30, Day 60, and Day 85.
Time Frame: Baseline, Day 30, Day 60, Day 85
Population: All participants who received study treatment
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Tiotropium | Revefenacin
Number analyzed (Participants) | 191 | 189
mL | 87 (15) | 78 (15)
Statistical Analysis 1: Comparison: Tiotropium vs Revefenacin; The OTE is defined as the average of the Day 30, Day 60, and Day 85 Revefenacin - Tiotropium Least Squares Mean differences. The null hypothesis was that the OTE Revefenacin - Tiotropium Least Squares Mean Difference was zero and the alternative hypothesis was that it was nonzero; Test type: Superiority; Mixed Models Analysis — The familywise type 1 error rate is controlled at 0.05 by testing the primary and secondary endpoint hypotheses in sequence and stopping after the first failure to reject the null hypothesis. Accordingly, the p-value is not shown; Mean Difference (Net) = -9, 95% CI 2-sided [-38 to 20] — Revefenacin - Tiotropium Least Squares Mean Difference; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: FEV1
Description: Change from baseline in FEV1 at trough on Day 30
Time Frame: Baseline, Day 30
Population: All participants who received study treatment
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Tiotropium | Revefenacin
Number analyzed (Participants) | 191 | 189
mL | 81 (16) | 83 (16)
Statistical Analysis 1: Comparison: Tiotropium vs Revefenacin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = 2, 95% CI 2-sided [-29 to 32] — Revefenacin - Tiotropium Least Squares Mean Difference; [other analysis details as in outcome 1, analysis 1]

4. Secondary Outcome: FEV1
Description: Change from baseline in FEV1 at trough on Day 60
Time Frame: Baseline, Day 60
Population: All participants who received study treatment
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Tiotropium | Revefenacin
Number analyzed (Participants) | 191 | 189
mL | 79 (17) | 73 (17)
Statistical Analysis 1: Comparison: Tiotropium vs Revefenacin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -6, 95% CI 2-sided [-40 to 29] — Revefenacin - Tiotropium Least Squares Mean Difference; [other analysis details as in outcome 1, analysis 1]

5. Secondary Outcome: FVC
Description: Change from baseline in forced vital capacity (FVC) at trough on Day 85
Time Frame: Baseline, Day 85
Population: All participants who received study treatment
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Tiotropium | Revefenacin
Number analyzed (Participants) | 191 | 189
mL | 198 (35) | 156 (35)
Statistical Analysis 1: Comparison: Tiotropium vs Revefenacin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -41, 95% CI 2-sided [-118 to 35] — Revefenacin - Tiotropium Least Squares Mean Difference; The Revefenacin - Tiotropium Least Squares Mean Difference was estimated by fitting a repeated measures mixed model which included terms for participant, treatment, 6 categorical covariates, and 3 continuous covariates: baseline FVC, screening FVC, and baseline PIFR. The 6 categorical covariates were reversibility to ipratropium status (reversible/not reversible), smoking status (current/former), concomitant LABA or LABA/ICS use (Yes/No), GOLD airflow category (3/4, i.e., postipratropium FEV1 % predicted < 30%/≥ 30%), sex (woman/man), and age group (< 65/≥ 65)

6. Secondary Outcome: 80-mL Increase in FEV1 at Trough on Day 85
Description: Participants with an 80-mL or greater change from baseline FEV1 at trough were counted as responders. Participants with change from baseline FEV1 < 80 mL and participants with change from baseline FEV1 not obtained were counted as nonresponders.
Time Frame: Baseline, Day 85
Population: All participants who received study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium | Revefenacin
Number analyzed (Participants) | 191 | 189
Participants | 83 | 63
Statistical Analysis 1: Comparison: Tiotropium vs Revefenacin; The null hypothesis was that the Revefenacin / Tiotropium responder Odds Ratio was equal to 1 and the alternative hypothesis was that it was not equal to 1; Test type: Superiority; Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.39 to 0.92] — The profile likelihood method was used to estimate the Revefenacin / Tiotropium responder OR; The Revefenacin / Tiotropium responder OR was estimated by fitting a logistic regression model which included terms for participant, treatment, 6 categorical covariates, and 3 continuous covariates: baseline FEV1, screening FEV1, and baseline PIFR. The 6 categorical covariates were reversibility to ipratropium status (reversible/not reversible), smoking status (current/former), concomitant LABA or LABA/ICS use (Yes/No), GOLD airflow category (3/4, i.e., postipratropium FEV1 % predicted < 30%/≥ 30%), sex (woman/man), and age group (< 65/≥ 65)

7. Secondary Outcome: First Occurrence of CompEx Event
Description: Count of participants experiencing events and time from first dose to first occurrence of a composite endpoint for exacerbations of COPD (CompEx) event were evaluated. The statistical analysis is a Cox proportional hazards model analysis of time to first event and the Revefenacin / Tiotropium hazard ratio is calculated and reported. Data are reported as the numbers of subjects with events and the hazard ratio is included in the Statistical Analysis section attached to the Outcome Measure data table.
  CompEx events are a composite of moderate or severe COPD exacerbation, premature termination from the study for any reason other than Sponsor decision, and clinically relevant deterioration in COPD. Clinically relevant deterioration events are defined as increases in COPD symptoms meeting specified criteria based on participant diary data.
Time Frame: Date of first dose through date of last dose + 7 days
Population: All participants who received study treatment and were evaluable for rescue medication use (i.e., were not using nebulized albuterol for rescue or albuterol 4 times daily for maintenance)
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium | Revefenacin
Number analyzed (Participants) | 174 | 176
Participants | 56 | 58
Statistical Analysis 1: Comparison: Tiotropium vs Revefenacin; The null hypothesis was that the Revefenacin / Tiotropium CompEx Event Hazard Ratio was equal to 1 and the alternative hypothesis was that it was not equal to 1; Test type: Superiority; Regression, Cox — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.69 to 1.45] — The profile likelihood method was used to estimate the Revefenacin / Tiotropium HR; The Revefenacin / Tiotropium HR was estimated by fitting a Cox proportional hazards model which included terms for participant, treatment, 6 categorical covariates, and 3 continuous covariates: baseline FEV1, screening FEV1, and baseline PIFR. The 6 categorical covariates were reversibility to ipratropium status (reversible/not reversible), smoking status (current/former), concomitant LABA or LABA/ICS use (Yes/No), GOLD airflow category (3/4, i.e., postipratropium FEV1 % predicted < 30%/≥ 30%), sex (woman/man), and age group (< 65/≥ 65)

ADVERSE EVENTS:
Time Frame: Day 1 through 7 days after the date of the last study drug dose.
Arm/Group | Tiotropium | Revefenacin
All-Cause Mortality (participants affected / at risk) | 0/191 | 0/189
Serious Adverse Events (participants affected / at risk) | 15/191 | 16/189
Other Adverse Events (participants affected / at risk) | 33/191 | 38/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium (N=191) | Revefenacin (N=189)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 3
Chronic left ventricular failure (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 2
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 2
Pneumonia legionella (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium (N=191) | Revefenacin (N=189)
Nausea (Gastrointestinal disorders) | 4 | 2
COVID-19 (Infections and infestations) | 1 | 3
Cellulitis (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Headache (Nervous system disorders) | 5 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 22 | 22 — Treatment-emergent COPD exacerbations were coded to this preferred term.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT05165485/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT05165485/SAP_001.pdf